CLINICAL TRIAL: NCT03403400
Title: "Can A Prescribed Walking Program With or Without Monitoring Impact Dizziness in the Older Adults?"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Adventist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1038487
Record Dates: First submitted 2017-12-29; First posted 2018-01-18 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Intervention Model Description: Experimental Design. To answer the study objective, a pragmatic, randomized, prospective, clinical study on 54 older adults with dizziness will be utilized. This will be conducted at Florida Hospital Sports Medicine and Rehabilitation locations that offer vestibular therapy. These are in East Orlando and Winter Park.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VRWP Group (Experimental): Vestibular Rehabilitation plus Walking with Pedometer Groupd
  Interventions: Behavioral: VRWP Group
- VRW Group (Active Comparator): Vestibular Rehabilitation plus Walking without Pedometer Group
  Interventions: Behavioral: VRW Group
- VR Group (No Intervention): Vestibular Rehabilitation Only Group. The VR (control) group will follow the conventional VR physical therapy without the encouragement of walking and without specification of walking in the home exercise program.

INTERVENTIONS:
Behavioral: VRWP Group — The VRWP group will have VR with an instruction to increase their number of steps daily to at least 3,000 steps using the pedometer (VR plus walking plus pedometer group). They will receive pedometers (Fitbit Zip), instructions on how to use the pedometer, step log forms, with home instruction handout to walk more at least more than ten minutes at a time. The participants will record on their activity log the number of steps shown on the step display at the end of the day. The daily step log form will be given to the research staff every visit for recording. The research staff will encourage their participants to increase their daily steps at least 10% until they achieve at least 3,000 steps daily.
  Arms: VRWP Group
Behavioral: VRW Group — The VR (control) group will follow the conventional VR physical therapy without the encouragement of walking and without specification of walking in the home exercise program.
  Arms: VRW Group

SUMMARY:
Dizziness is a common complaint reported by 30% of people above 65 years of age and by more than 50% of those 90 years of age and older.(1) Age-related decline in vestibular, musculoskeletal, and neurologic performances compounded by a vestibular pathology can result to debilitating physical and psychological consequences. Dizziness is associated with falls,(2) disability (3) and physical inactivity.(4) Walking for endurance is cited as one of the components of vestibular rehabilitation (VR) in the "Clinical Practice Guideline for Peripheral Vestibular Hypofunction".(5) Although walking can offset the avoidance of physical activity from symptom provocation, no direct evidence has been found to support the effect of walking on postural and dynamic stability, function, and participation in people with dizziness.

The primary purpose of this study is to evaluate the impact of walking as an exercise component of VR on both primary and secondary vestibular-specific outcome measures. The primary outcomes are mCTSIB, TUG test, DGI, and DHI, while the secondary outcomes are the total number of visits and length of interventions (in weeks). The second purpose is to evaluate whether pedometers increase the adherence of older adults with vestibular issues to a walking program. This will be measured by change in physical activity, as represented by International Physical Activity Questionnaire (IPAQ) Walking Metabolic Equivalent of Task (MET)-minutes/week and IPAQ Total Physical Activity MET-minutes/week scores from the IPAQ short form during the episode of care (admission and discharge) and on four-weeks follow-up compared to those patients who only received instructions to walk without a pedometer. The third purpose of this study is to establish test-retest reliability of the TUG test on older adults with dizziness. Lastly, the fourth purpose of this study to investigate if the TUG, DGI, and mCTSIB are significant and strong predictors of the DHI in older adults with dizziness. Protocol #1365169 "Predictors of Disability in the Older Adults" is being performed to supplement the number of subjects for the fourth objective of this study.

DETAILED DESCRIPTION:
Research Design

1. Experimental Design. To answer the first and second study objectives, a pragmatic, randomized, prospective, clinical study on 54 older adults with dizziness will be utilized. This will be conducted at Florida Hospital Sports Medicine and Rehabilitation locations that offer vestibular therapy. These are in East Orlando and Winter Park.
2. Correlation Design. A correlation analysis will be performed on the data collected on 54 subjects in the experimental design to establish the test-retest reliability of the Timed Up and Go.
3. Cross-sectional Descriptive Design. A regression analysis will be performed on three predictors of the Dizziness Handicap Inventory, obtained from the data collected on 54 subjects in the experimental design and from Florida Hospital Sports Medicine and Rehabilitation Physical Therapy medical charts from June 2015 to June 2018 that met the inclusion and exclusion criteria that were outlined in the Protocol #1365169.

For the experimental design that will be conducted at Florida Hospital locations, the following data will be collected as standard of care by the physical therapist during initial evaluation, and if more time is needed, during the first follow-up physical therapy appointment: mCTSIB, TUG, DGI, DHI, age, gender, body mass index, home situation, Functional Comorbidity Index (FCI) total, ability to drive, medications and insurance type. After the subject signs the informed consent prior to the tenth visit, the study coordinator will be notified by the research staff to conduct a retrospective chart review of the patient's medical record. The study coordinator will extract the following baseline measurements from the subject's medical record: DGI, mCTSIB, DHI, TUG and socio-demographic data that include age, gender, body mass index, home situation (lives alone or with social support), Functional Comorbidity Index (FCI) total, ability to drive (able or unable), medications for vertigo and insurance type (Medicare/Non-medicare). Based on the retrospective chart review, the study coordinator will determine if the subject is eligible to participate in the study.

Visit 1: Once the study coordinator determined that the subject is eligible to participate in the study, the subject will be assigned a research number and will be randomized into one of the three intervention groups. The research staff can initiate or continue the VR program and initiate the research intervention according to the intervention group. For the test-retest reliability of the TUG test, there will be one practice trial followed by two final performances that will be included in the data analysis. The subject will also be asked to complete the IPAQ-short form questionnaire. The test-retest reliability of TUG and the IPAQ-short form questionnaire are for research purposes only.

Visit 2: The research staff can initiate the research intervention according to the intervention group.

Visit 3 to visit prior to discharge: The research staff can continue the VR and intervention according to the intervention group.

Discharge or last visit: All outcome measures (DGI, TUG, mCTSIB, DHI and IPAQ) will be reassessed. Discharge scores for DGI, TUG, mCTSIB and DHI are standard of care, while IPAQ is for research purposes only. The total number of visits and length of interventions (in weeks) for every participant will be recorded as secondary outcome measures. These research data will be forwarded to the study coordinator, and will be stored in a locked cabinet and password protected Florida Hospital computer.

Four-weeks after discharge: The study coordinator will conduct a follow up phone call to all subjects four weeks after discharge summary is completed to obtain the level of physical activity using the IPAQ short form questionnaire. This is for research purposes only. A follow-up on a subject will be discontinued if a subject is not reached after three attempts of follow-up phone call made on three different days between 30 and 45 days. Data analysis will commence once all the data from 54 subjects are collected.

Sample Size Determination

A priori power analysis predicting a large effect size (F=.25) determined that a total of 54 subjects (18 in each group), who met the inclusion and exclusion criteria will be needed, with alpha at the conventional value of .05 to achieve a .80 power, that includes an assumption of a dropout rate of 50% .

Statistical Analysis Plan

The results will be presented through the following tables with supporting explanations:

* Clinical and sociodemographic characteristics of participants by group at baseline.
* Comparisons of TUG, DGI, mCTSIB and DHI between the three intervention groups on admission and discharge.
* Comparisons of self-reported walking activity (walking MET-min/week) and total self-reported energy expenditure (total physical activity MET-min/week) as determined from the IPAQ short form on admission, discharge and four-week follow-up between the three intervention groups
* Comparisons of averages of compliance to step log recording and compliance rate for meeting step goal between the VRWP and VRW groups. Compliance is defined as low (<33%), moderate (33%-75%) and high (>75%) based on the step log or walking log. This grading of compliance was used by Hall and colleagues in their research on efficacy of gaze stability exercises in older adults with dizziness.(6)
* Comparisons of total number of visits and length of interventions in weeks between the three intervention group.
* Intraclass Correlation Coefficients for the Timed Up and Go test-retest reliability
* Result of stepwise linear regression analysis for TUG, DGI, mCTSIB and DHI

All interval and ratio data will be tested for normality prior to undertaking the data analysis. Descriptive statistics will be used to describe the characteristics of the sample and compare the three groups at baseline. This will include Analysis of Variance (ANOVA) for parametric and Chi Square for nonparametric sociodemographic and clinical data.

Analyses will employ five repeated measures Analysis of Covariance (ANCOVA), adjusting for age, with two independent variables (group and time) and five outcome measures (TUG, DGI, DHI, mCTSIB and IPAQ short form). The adjustment of age is based on age-related decline. Intraclass Correlation Coefficient will be calculated to establish the test-retest reliability of the TUG and a stepwise linear regression with age as covariant will be conducted for all 54 subjects at baseline to determine if TUG, mCTSIB and DGI are predictors of DHI. Two-tailed test will be utilized to compare the compliance with step log recording and meeting step goals between the two walking groups (VRWP and VRW), and ANOVA to compare of total number of visits and total length of intervention in weeks between the three groups. Alpha for all analyses will be set at 0.05 to test for significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older referred for physical therapy evaluation for symptoms of dizziness, postural instability, or both
2. Able to walk without the physical help of another person, with or with no assistive device
3. Able to follow commands and execute the examination and intervention instructions in the English language
4. Willing to participate in a phone interview four weeks after discharge
5. Able to provide informed consent

Exclusion Criteria:

1. Unstable medical issues, such as unstable or uncontrolled cardiovascular conditions, elevated blood pressure (Systolic greater than or equal to 140mmHg and diastolic greater than or equal to 90mmHg), orthostatic hypotension (a fall in systolic blood pressure of at least 20mmHg or diastolic blood pressure of at least 10mmHg when a person stands from a sitting or lying down position), uncontrolled metabolic disease, as determined by the evaluating physical therapist, documented in the Functional Comorbidity Index, vital signs and assessment portion of the initial evaluation.
2. History of falls from syncopal origin
3. Dizziness of central origin, such as stroke, head injuries, MS or PD;
4. Active BPPV (patients with positive dix hallpike and/or roll test)
5. Inability to walk without physical assistance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Blackinton, EED, Study Director — Nova Southeastern University; Joann Gallichio, DSC, Study Director — Nova Southeastern University; Ann Galgon, PhD, Study Director — University of the Sciences; Leana Araujo, PhD, Study Director — Adventist University
Locations (2):
- United States (2):
  - Florida Hospital East Orlando, Orlando, Florida
  - Florida Hospital Winter Park, Winter Park, Florida

REFERENCES:
- [Background] Maarsingh OR, Stam H, van de Ven PM, van Schoor NM, Ridd MJ, van der Wouden JC. Predictors of dizziness in older persons: a 10-year prospective cohort study in the community. BMC Geriatr. 2014 Dec 15;14:133. doi: 10.1186/1471-2318-14-133. PMID 25510936
- [Background] Liston MB, Bamiou DE, Martin F, Hopper A, Koohi N, Luxon L, Pavlou M. Peripheral vestibular dysfunction is prevalent in older adults experiencing multiple non-syncopal falls versus age-matched non-fallers: a pilot study. Age Ageing. 2014 Jan;43(1):38-43. doi: 10.1093/ageing/aft129. Epub 2013 Sep 15. PMID 24042003
- [Background] Mueller M, Strobl R, Jahn K, Linkohr B, Ladwig KH, Mielck A, Grill E. Impact of vertigo and dizziness on self-perceived participation and autonomy in older adults: results from the KORA-Age study. Qual Life Res. 2014 Oct;23(8):2301-8. doi: 10.1007/s11136-014-0684-x. Epub 2014 Apr 10. PMID 24719016
- [Background] Mueller M, Strobl R, Jahn K, Linkohr B, Peters A, Grill E. Burden of disability attributable to vertigo and dizziness in the aged: results from the KORA-Age study. Eur J Public Health. 2014 Oct;24(5):802-7. doi: 10.1093/eurpub/ckt171. Epub 2013 Nov 8. PMID 24213583
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Background] Hall CD, Heusel-Gillig L, Tusa RJ, Herdman SJ. Efficacy of gaze stability exercises in older adults with dizziness. J Neurol Phys Ther. 2010 Jun;34(2):64-9. doi: 10.1097/NPT.0b013e3181dde6d8. PMID 20588090
- [Background] Horn LB, Rice T, Stoskus JL, Lambert KH, Dannenbaum E, Scherer MR. Measurement Characteristics and Clinical Utility of the Clinical Test of Sensory Interaction on Balance (CTSIB) and Modified CTSIB in Individuals With Vestibular Dysfunction. Arch Phys Med Rehabil. 2015 Sep;96(9):1747-8. doi: 10.1016/j.apmr.2015.04.003. No abstract available. PMID 26550644
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Whitney SL, Marchetti GF, Schade A, Wrisley DM. The sensitivity and specificity of the Timed "Up & Go" and the Dynamic Gait Index for self-reported falls in persons with vestibular disorders. J Vestib Res. 2004;14(5):397-409. PMID 15598995
- [Background] Wrisley DM, Walker ML, Echternach JL, Strasnick B. Reliability of the dynamic gait index in people with vestibular disorders. Arch Phys Med Rehabil. 2003 Oct;84(10):1528-33. doi: 10.1016/s0003-9993(03)00274-0. PMID 14586922
- [Background] Shumway-Cook A, Baldwin M, Polissar NL, Gruber W. Predicting the probability for falls in community-dwelling older adults. Phys Ther. 1997 Aug;77(8):812-9. doi: 10.1093/ptj/77.8.812. PMID 9256869
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Shook RP, Gribben NC, Hand GA, Paluch AE, Welk GJ, Jakicic JM, Hutto B, Burgess S, Blair SN. Subjective Estimation of Physical Activity Using the International Physical Activity Questionnaire Varies by Fitness Level. J Phys Act Health. 2016 Jan;13(1):79-86. doi: 10.1123/jpah.2014-0543. Epub 2015 Apr 21. PMID 25898394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited from July 2018 - September 2019 through consecutive admissions from two outpatient clinics with therapists with experience in VR.
Pre-assignment Details: After the subject signed the informed consent, the study coordinator was notified by the research staff to conduct a retrospective chart review of the medical record of the subject. Based on the retrospective chart review, the study coordinator determined if the subject was eligible to participate in the study.
Period: Overall Study
Arm/Group | VRWP Group | VRW Group | VR Group
Started | 5 | 6 | 6
Completed | 3 | 6 | 4
Not Completed | 2 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Hospitalization | 1 | 0 | 0
Not completed — Benign Paroxysmal Positional Vertigo | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRWP Group | VRW Group | VR Group | Total
Number analyzed (Participants) | 3 | 6 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.67 (10.41) | 81.17 (9.81) | 78.25 (8.81) | 79.03 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 4 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
IPAQ-Walk [Mean (Standard Deviation); unit: METS-min/week] | 660 (646.03) | 562.07 (212.10) | 2293.5 (4020.56) | 1171.86 (1626.23)
IPAQ-Total [Mean (Standard Deviation); unit: METS-min/week] | 1046.67 (805.75) | 2145.4 (2667.75) | 3963.5 (6573.74) | 2385.19 (3349.08)

OUTCOME MEASURES:

1. Primary Outcome: Modified Clinical Test of Sensory Integration for Balance (mCTSIB)
Description: The mCTSIB quantifies the ability of the patient to use information from somatosensory, visual and vestibular system effectively for postural stability. This test eliminated conditions 3 and 6 of the original CTSIB, which use an altered visual input (visual conflict dome). It is performed with the feet together, a modification from the original test, which is with feet apart.(7) The four conditions of mCTSIB are standing on firm surface eyes open, standing on firm surface eyes closed, standing on compliant surface eyes open, and standing on compliant surface eyes closed. The patient is timed for 30 seconds and the average score of three trials is obtained. It only requires a timer and balance foam to administer the test.
Time Frame: Change from up to week 9 of treatment to up to 16 weeks of treatment
Population: Pretest and posttest means of VR (n=5), VRWP (n=4) and VRW (n=6) were presented. Another arm was added combining VRWP and VRW data into a group representing prescribed walking (n=10)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Control (VR) Group: Vestibular Rehabilitation Only Group. The VR (control) group will follow the conventional VR physical therapy without the encouragement of walking and without specification of walking in the home exercise program.
- VRWP (Vestibular Rehabilitation With Walking With Pedometer): Vestibular Rehabilitation with Walking with Pedometer. The VRWP group (N=4) had VR with an instruction to increase their number of steps daily to at least 3,000 steps using the pedometer (VR plus walking plus pedometer group).
- VRW (Vestibular Rehabilitation Walking Without a Pedometer): Vestibular Rehabilitation with Walking without a Pedometer. The VRW group (N=6) received VR and a time-based instruction to walk more daily at least 10 minutes at a time (VR plus walking no pedometer group).
- Prescribed Walking Group: VRWP and VRW data were combined into a group representing prescribed walking.
Arm/Group | Control (VR) Group | VRWP (Vestibular Rehabilitation With Walking With Pedometer) | VRW (Vestibular Rehabilitation Walking Without a Pedometer) | Prescribed Walking Group
Number analyzed (Participants) | 5 | 4 | 6 | 10
seconds
  Pretest | 115.98 (5.82) | 97.4 (5.78) | 110.15 (9.97) | 107.23 (10.55)
  Posttest | 120 (0) | 111.17 (10.234) | 118 (3.35) | 115.27 (7.23)
Statistical Analysis 1: Comparison: Control (VR) Group vs VRWP (Vestibular Rehabilitation With Walking With Pedometer) vs VRW (Vestibular Rehabilitation Walking Without a Pedometer); Ho: There is no significant difference between groups in mCTSIB Ha: There is a significant difference between groups in mCTSIB; Test type: Equivalence — Comparison of variance; p = .640, Kruskal-Wallis; Test Statistics = .893
Statistical Analysis 2: Comparison: Control (VR) Group vs Prescribed Walking Group; Ho: There is no significant difference between the prescribed walking group and the control group in mCTSIB Ha: There is a significant difference between the prescribed walking group and the control group in mCTSIB; Test type: Equivalence — Comparison of variance; p = .18, Kruskal-Wallis; Test Statistics = .196

2. Primary Outcome: Timed Up and Go (TUG) Test
Description: The TUG is a test of balance and risk for falls.(8) This test measures the time it takes to walk 3 meters starting from a sitting position and it ends when the patient is seated again. Among the population studied for the TUG are the frail elderly and vestibular disorders.(9) The cut-off scores that indicate risk for falls are greater than 13.5 seconds for community dwelling older adults (8) and greater than 11.1 seconds for vestibular disorders.(10)
Time Frame: Change from up to week 9 of treatment to up to 16 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Vestibular Rehabilitation With Walking With Pedometer (VRWP): The VRWP group (N=4) had VR with an instruction to increase their number of steps daily to at least 3,000 steps using the pedometer (VR plus walking plus pedometer groupVestibular Rehabilitation with Walking without a Pedometer.
- Vestibular Rehabilitation Walking Without a Pedometer (VRW): The VRW group (N=6) received VR and a time-based instruction to walk more daily at least 10 minutes at a time (VR plus walking no pedometer group).
- Prescribed Walking (VRWP +VRW) Group: The Prescribed Walking group is composed of 4 subjects walking with pedometer (VRWP) and 6 subjects walking without pedometer (VRW).
Arm/Group | Control (VR) Group | Vestibular Rehabilitation With Walking With Pedometer (VRWP) | Vestibular Rehabilitation Walking Without a Pedometer (VRW) | Prescribed Walking (VRWP +VRW) Group
Number analyzed (Participants) | 5 | 4 | 6 | 10
seconds
  Pretest | 10 (1.64) | 12.73 (3.54) | 12.42 (5.75) | 12.54 (4.75)
  Posttest | 7.80 (1.3) | 10 (3.46) | 10.92 (5.12) | 10.55 (4.34)
Statistical Analysis 1: Comparison: Control (VR) Group vs Vestibular Rehabilitation With Walking With Pedometer (VRWP) vs Vestibular Rehabilitation Walking Without a Pedometer (VRW); Ho: There is no significant difference between the groups in TUG Ha: There is a significant difference between the groups in TUG; Test type: Equivalence — comparison of variance; p = .67, Kruskal-Wallis; Test Statistics = .803
Statistical Analysis 2: Comparison: Control (VR) Group vs Prescribed Walking (VRWP +VRW) Group; Ho: There is no significant difference in TUG between the prescribed walking and control group Ha: There is a significant difference in TUG between the prescribed walking and control group; Test type: Equivalence — comparison of variance; p = .71, Kruskal-Wallis; Test Statistics = .14

3. Primary Outcome: Dynamic Gait Index
Description: The DGI assesses the ability to maintain balance while walking in the presence of external demands. It is scored based on a 4-point ordinal scale (3=no gait dysfunction, 2=minimal impairment, 1=moderate impairment and 0=severe impairment) with the highest possible score of 24.(11) A cut-off score of less than 19 is indicative of increased fall risks in community-dwelling elderlies.(12)
Time Frame: Change from up to week 9 of treatment to up to 16 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Groups:
- Vestibular Rehabilitation With Walking With Pedometer: The VRWP group (N=4) had VR with an instruction to increase their number of steps daily to at least 3,000 steps using the pedometer (VR plus walking plus pedometer groupVestibular Rehabilitation with Walking without a Pedometer.
- Vestibular Rehabilitation Walking Without Pedometer (VRW): The VRW group (N=6) received VR and a time-based instruction to walk more daily at least 10 minutes at a time (VR plus walking no pedometer group).
- Prescribed Walking (VRWP +VRW) Group: The walking group is composed of the VRWP (Vestibular Rehabilitation with Walking with Pedometer) and VRW (Vestibular Rehabilitation with Walking without Pedometer
Arm/Group | Control (VR) Group | Vestibular Rehabilitation With Walking With Pedometer | Vestibular Rehabilitation Walking Without Pedometer (VRW) | Prescribed Walking (VRWP +VRW) Group
Number analyzed (Participants) | 5 | 4 | 6 | 10
score
  Pretest | 20 (2.74) | 19.5 (2.38) | 20.67 (2.88) | 20.2 (2.62)
  Posttest | 22.80 (1.64) | 22 (1.63) | 22.67 (1.03) | 22.4 (1.26)
Statistical Analysis 1: Comparison: Control (VR) Group vs Vestibular Rehabilitation With Walking With Pedometer vs Vestibular Rehabilitation Walking Without Pedometer (VRW); Ho: There is no significant difference between the groups in DGI Ha: There is a significant difference between the groups in DGI; Test type: Equivalence — Comparison of variance; p = .67, Kruskal-Wallis; Test Statistics = .803, Standard Deviation 1.79
Statistical Analysis 2: Comparison: Control (VR) Group vs Prescribed Walking (VRWP +VRW) Group; Ho: There is no significant difference between the prescribed walking group and the control group in DGI Ha: There is a significant difference between the prescribed walking group and control group in DGI; Test type: Equivalence — comparison of variance; p = .42, Kruskal-Wallis; Test Statistics = .66

4. Primary Outcome: Dizziness Handicap Inventory (DHI)
Description: The DHI is a 25-item self-report questionnaire that quantifies the functional, emotional and physical impact of dizziness. Answers are graded 0 for no, 2 for sometimes and 4 for yes, with a maximum total score of 100. Interpretations are mild dizziness for scores between 0-30, moderate for 31-60 and severe for 61-100.(13)
Time Frame: Change from up to week 9 of treatment to up to 16 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Groups:
- Prescribed Walking Group (VRWP+VRW): The walking group is composed of the VRWP (Vestibular Rehabilitation with Walking with Pedometer) and VRW (Vestibular Rehabilitation with Walking without Pedometer)
Arm/Group | Control (VR) Group | Vestibular Rehabilitation With Walking With Pedometer | Vestibular Rehabilitation Walking Without Pedometer (VRW) | Prescribed Walking Group (VRWP+VRW)
Number analyzed (Participants) | 5 | 4 | 6 | 10
score
  Pretest | 16 (22.56) | 38.5 (31.09) | 23.67 (13.65) | 29.6 (22.01)
  Posttest | 13.2 (18.9) | 11.5 (9.71) | 7.33 (5.16) | 9 (7.13)
Statistical Analysis 1: Comparison: Control (VR) Group vs Vestibular Rehabilitation With Walking With Pedometer vs Vestibular Rehabilitation Walking Without Pedometer (VRW); Ho: There is no significant difference between the groups in DHI Ha: There is a significant difference between the groups in DHI; Test type: Equivalence — comparison of variance; p = .11, Kruskal-Wallis; Test Statistics = 4.386
Statistical Analysis 2: Comparison: Control (VR) Group vs Prescribed Walking Group (VRWP+VRW); Ho: There is no significant difference in DHI between the prescribed walking group and the control group Ha: There is a significant difference in DHI between the prescribed walking group and the control group; Test type: Equivalence — comparison of variance; p = .04, Kruskal-Wallis; Test Statistics = 4.351

5. Secondary Outcome: Total Number of Visits
Description: The total number of visits after signing the informed consent between the three intervention groups were compared.
Time Frame: From initial evaluation (day 1 of treatment) to up to 16 weeks of treatment
Population: There are 5 participants in the Control (Vestibular Rehabilitation) Group and 10 Walking Group. Participants in the Walking Group received a prescribed walking program in the form of pedometer (Vestibular Rehabilitation plus walking with pedometer or VRWP N=4 and timed-walking (Vestibular Rehabilitation plus walking without Pedometer or VRW N=6).
Measure: Mean (Standard Deviation); unit: visits
Groups:
- Vestibular Rehabilitation Walking With no Pedometer (VRW): The VRW group (N=6) received VR and a time-based instruction to walk more daily at least 10 minutes at a time (VR plus walking no pedometer group).
- Prescribed Walking (VRWP +VRW) Group: The Prescribed walking group is composed of the VRWP (Vestibular Rehabilitation with Walking with Pedometer) and VRW (Vestibular Rehabilitation with Walking without Pedometer
Arm/Group | VR Group | Vestibular Rehabilitation With Walking With Pedometer (VRWP) | Vestibular Rehabilitation Walking With no Pedometer (VRW) | Prescribed Walking (VRWP +VRW) Group
Number analyzed (Participants) | 5 | 4 | 6 | 10
visits | 5.6 (1.03) | 6.75 (1.89) | 7.33 (1.89) | 7.04 (1.89)

6. Secondary Outcome: Length of Interventions in Weeks
Description: The length of interventions in weeks between the three intervention group will be compared.
Time Frame: From initial evaluation (day 1 of treatment) to up to 16 weeks of treatment
Population: Means and Standard Deviations of VR (n=5), VRWP (n=4) and VRW (n=6) were presented. Another arm was added combining VRWP and VRW data into a group representing prescribed walking (n=10)
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Vestibular Rehabilitation With Walking With Pedometer (VRWP): The VRWP group (N=6) had VR with an instruction to increase their number of steps daily to at least 3,000 steps using the pedometer (VR plus walking plus pedometer groupVestibular Rehabilitation with Walking without a Pedometer.
Arm/Group | VR Group | Vestibular Rehabilitation With Walking With Pedometer (VRWP) | Vestibular Rehabilitation Walking With no Pedometer (VRW) | Prescribed Walking (VRWP +VRW) Group
Number analyzed (Participants) | 5 | 4 | 6 | 10
weeks | 8.5 (1.41) | 9.25 (1.65) | 8.5 (1.98) | 8.88 (1.82)

7. Other Pre Specified Outcome: International Physical Activity Questionnaire (IPAQ)- Walk
Description: The IPAQ short form is an instrument evaluation tool of physical activity among the adults. It has three categories: low, moderate and high. The specific type of activities assessed are walking, moderate intensity activities and vigorous intensity activities. All continuous scores are expressed in MET-minutes/week with walking =3.3 METs, Moderate PA=4.0 METs and Vigorous PA = 8.0 METs. An overall total physical activity score can be computed as the sum of the total MET-minutes/week scores.(14)
Time Frame: Change from up to week 9 of treatment to up to 4 weeks post treatment
Population: IPAQ-Walk scores were categorized as increase if there was an increase in four-weeks follow-up score compared to pretest score, same if there was no change in four-weeks follow-up score compared to pretest score, and decrease if there was a decline in four-weeks follow-up score compared to pretest score.
Measure: Number; unit: participants
Arm/Group | VRWP Group | VRW Group | VR Group
Number analyzed (Participants) | 3 | 6 | 4
participants
  increase | 3 | 4 | 2
  same | 0 | 0 | 0
  decrease | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | VRWP Group | VRW Group | VR Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Small sample size, lack of blinding, lack of intention-to-treat, lack of objective measures for physical activity, unequal distribution of subjects based on DHI severity score, retrospective data collection for predictors of DHI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT03403400/Prot_SAP_000.pdf